CLINICAL TRIAL: NCT04708951
Title: A Prospective Randomized Comparison of Colonoscopy Adenoma Detection Rate With a Disposable Cap (ENDOCUFF VISION®) (Endocuff) Versus a Permanently Mounted Balloon (G-EYE®)
Brief Title: Comparison of Adenoma Detection Rate With ENDOCUFF VISION® vs. G-EYE®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Horst Schmidt Klinik GmbH (Industry)
Responsible Party: Principal Investigator, Prof. Dr. Ralf Kiesslich, Prof., Dr. Horst Schmidt Klinik GmbH
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: ENDOCUFF vs. G-EYE
Record Dates: First submitted 2021-01-11; First posted 2021-01-14 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Adenoma; Colorectal Cancer
Keywords: Adenoma; Colorectal Cancer
MeSH Terms: conditions — Adenoma; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to one of two groups - ECV colonoscopy or G-EYE® colonoscopy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- ECV colonoscopy (Active Comparator): EndoCuff Vision® device (ECV)
  Interventions: Device: ENDOCUFF VISION® device
- G-EYE® colonoscopy (Experimental): G-EYE® colonoscope (G-EYE)
  Interventions: Device: G-EYE® colonoscope

INTERVENTIONS:
Device: ENDOCUFF VISION® device — ENDOCUFF VISION® is a disposable cap placed on the tip of a standard colonoscope, intended to flatten colonic folds and assist in controlling the colonoscope's field of view and tip positioning
  Arms: ECV colonoscopy
Device: G-EYE® colonoscope — The G-EYE® balloon is a reusable (reprocessable) balloon permanently installed on the distal tip of a standard colonoscope, and is also intended to assist in flattening colonic folds and control the colonoscope's field of view and tip positioning
  Arms: G-EYE® colonoscopy

SUMMARY:
The study is intended to compare the detection rate obtained by performing G-EYE® high definition colonoscopy vs. the detection rate obtained by performing ECV high definition colonoscopy.

DETAILED DESCRIPTION:
This is a multicenter, two-arm, randomized, open-label study intended to compare the detection rate obtained by performing G-EYE® high definition colonoscopy vs. the detection rate obtained by performing ECV high definition colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Screening and surveillance population for Adenoma and CRC.
2. The patient must understand and sign a written informed consent for the procedure.

Exclusion Criteria:

1. Subjects with inflammatory bowel disease;
2. Subjects with a personal history of hereditary polyposis syndrome;
3. Subjects with suspected chronic stricture potentially precluding complete colonoscopy;
4. Subjects with diverticulitis or toxic megacolon;
5. Subjects with prior colonic surgery (exclusion appendectomy)
6. Subjects with a history of radiation therapy to abdomen or pelvis;
7. Pregnant or lactating female subjects;
8. Subjects who are currently enrolled in another clinical investigation.
9. Subjects with current oral or parenteral use of anticoagulants, not considered eligible by the investigator.
10. Subjects with recent (within the last 3 mounts) coronary ischemia or CVA (stroke)
11. Any patient condition deemed too risky for the study by the investigator

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 970 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Comparison between adenoma detection rate of G-EYE® colonoscopy and EndoCuff Vision® | June 2021
  G-EYE® colonoscopy adenoma detection rate will be compared to the adenoma detection rate of EndoCuff Vision® colonoscopy. The primary performance measure is the adenoma detection rate (ADR), which is defined as the percentage of subjects with at least one adenoma found, in each of the study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Kiesslich, Prof., Principal Investigator — Helios Dr. Horst Schmidt Kliniken Wiesbaden
Locations (3):
- United States (2):
  - IU Health University Hospital, Indianapolis, Indiana
  - NYU Langone Health, New York, New York
- Helios Dr. Horst Schmidt Kliniken Wiesbaden, Wiesbaden, Germany

IPD SHARING:
Plan to Share IPD: No